CLINICAL TRIAL: NCT04710082
Title: Outcomes of a New Trans-epithelial Photorefractive Keratectomy (Streamlight PRK) Compared to Conventional PRK Procedures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mahmoud Abdel-Radi, Principal Investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TEPRK
Record Dates: First submitted 2021-01-08; First posted 2021-01-14 (Actual); Last update posted 2021-07-20 (Actual); Status verified 2021-07

CONDITIONS: Myopia ≤ -6 Diopters or Myopic Astigmatism ≤ -4 Diopters
Keywords: Photorefractive Keratectomy PRK; Phototherapeutic Keratectomy PTK; Trans-epithelial PRK; Laser Vision Correction LVC
MeSH Terms: interventions — Photorefractive Keratectomy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients planned to undergo conventional 2 step trans-epithelial PTK-PRK (Active Comparator): Patients planned to undergo:
  1. Epithelial removal using Phototherapeutic Keratectomy PTK as a separate step.
  2. Laser Vision Correction using Excimer laser wavefront optimized technology.
  Interventions: Procedure: Photorefractive keratectomy (PRK)
- Patients planned to undergo the new single step trans-epithelial (StreamLight) PRK. (Active Comparator): Patients planned to undergo:
  Epithelial removal and Excimer wavefront optimized Laser Vision Correction in a single step using the new StreamLight Technology.
  Interventions: Procedure: Photorefractive keratectomy (PRK)

INTERVENTIONS:
Procedure: Photorefractive keratectomy (PRK) — Photorefractive keratectomy (PRK) is a surgical procedure used by ophthalmic surgeons to treat patients presented with refractive errors and involves corneal epithelial removal followed by application of excimer laser to correct different refractive errors including Myopia, Hyperopia and Astigmatism.

SUMMARY:
Photorefractive keratectomy (PRK) involves mechanical or alcohol assisted debridement of the epithelium that leads to potential basement membrane (BM) injury ,with resultant more significant haze and pain compared to laser assisted epithelial removal known as 2 step trans-epithelial PRK (PTK-PRK). Our study is focusing on comparing the outcomes of the conventional 2 step trans-epithelial PTK-PRK to the new single step trans-epithelial PRK (StreamLight PRK, Alcon lab, TX, USA).

DETAILED DESCRIPTION:
Photorefractive keratectomy (PRK) is nowadays one of the commonest refractive procedures in laser vision correction (LVC). PRK differs from laser in situ keratomileusis (LASIK) in that it's a flapless procedure involving the removal of corneal epithelium with different techniques including manual removal , alcohol assisted removal or excimer laser assisted removal with phototherapeutic keratectomy (PTK). Mechanical or alcohol assisted debridement of the epithelium may lead to potential basement membrane (BM) injury ,with resultant more significant haze and pain compared to laser assisted epithelial removal known as 2 step trans-epithelial PRK (PTK-PRK).

Single step trans-epithelial PRK allows removing the epithelium and stroma in a single step with a single ablation profile.

Previous studies paid particular attention for comparing the 2 step PTK-PRK procedure or the new single step PRK procedure to the conventional PRK procedures involving epithelial removal whether manual or alcohol assisted.

The aim of this study is to focus on comparing the different outcomes of the new single step Trans-epithelial PRK (StreamLight Technology) versus the routine 2 step PTK-PRK in terms of postoperative vision, epithelial healing, pain scoring and haze evaluation.

ELIGIBILITY:
* Inclusion Criteria: Candidates for Laser vision correction (LVC) with

  1. Myopia up to -6 diopters
  2. Myopic astigmatism up to -4 diopters
  3. Corneal thinnest location ≥ 500 um and a residual stromal bed ≥ 300um.
* Exclusion criteria

  1. Patients not candidates for LVC.
  2. Hyperopic patients.
  3. Systemic disease that contraindicates LVC.
  4. Intra- or post-operative complications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Uncorrected distant visual acuity (UDVA) | 6 months
  Visual acuity measurement using Snellen's Acuity Chart and will be expressed as decimal notation
Postoperative Refraction (Spherical equivalent) | 6 months
  Measured by Topcon Auto-Keratorefractometer

SECONDARY OUTCOMES:
Epithelial healing duration | 2 weeks
  Time for the epithelium to heal reported in days after PRK procudre
Postoperative pain | 1 week
  Verbal Rating Scale(a series of words commonly used to describe pain (0: no pain, 1: mild pain, 2: moderate pain, 3: severe pain, 4: disabling pain)
Postoperative Haze | 3 months
  Corneal Haze scoring using slit lamp bio-microscopy according to Fantes scoring system:
  0: No haze, completely clear cornea
  0.5: Trace haze seen with careful oblique illumination
  1. Haze not interfering with visibility of fine iris details
  2. Mild obscuration of iris details
  3. Moderate obscuration of the iris and lens
  4. Complete opacification of the stroma in the area of the scar, anterior chamber is totally obscured

CONTACTS AND LOCATIONS:
Locations (1):
- TIBA eye center, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kaluzny BJ, Cieslinska I, Mosquera SA, Verma S. Single-Step Transepithelial PRK vs Alcohol-Assisted PRK in Myopia and Compound Myopic Astigmatism Correction. Medicine (Baltimore). 2016 Feb;95(6):e1993. doi: 10.1097/MD.0000000000001993. PMID 26871764
- [Derived] Abdel-Radi M, Shehata M, Mostafa MM, Aly MOM. Transepithelial photorefractive keratectomy: a prospective randomized comparative study between the two-step and the single-step techniques. Eye (Lond). 2023 Jun;37(8):1545-1552. doi: 10.1038/s41433-022-02174-4. Epub 2022 Jul 21. PMID 35864163